CLINICAL TRIAL: NCT07223242
Title: Tailored Exercise Training Study Among Adults With HFpEF
Acronym: TEXPEF
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Ambarish Pandey, Associate Professor of Medicine, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STU-2024-0592
Record Dates: First submitted 2025-10-06; First posted 2025-10-31 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-10

CONDITIONS: HFpEF - Heart Failure With Preserved Ejection Fraction; Diabetic Cardiomyopathies
Keywords: Diabetic cardiomyopathy; Remote exercise training; Weight loss; Rehab
MeSH Terms: conditions — Diabetic Cardiomyopathies; Weight Loss | interventions — Resistance Training

STUDY DESIGN:
Intervention Model Description: Participants will be randomized in a 1:1:1:1 fashion for phase 2
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Moderate-intensity continuous training (MCT) (Active Comparator): Tailored moderate-intensity exercise training video with weekly virtual meetings with a coach
  Interventions: Behavioral: Moderate-intensity continuous training (MCT)
- Moderate-intensity continuous training + weight loss (Experimental): Tailored moderate-intensity exercise training videos with weekly virtual meetings with a coach + initiation/intensification of pharmacological weight loss
  Interventions: Behavioral: Moderate-intensity continuous training (MCT); Drug: Weight loss
- Moderate-intensity continuous training + resistance training (Experimental): Tailored moderate-intensity exercise training videos with weekly virtual meetings with a coach + tailored resistance training videos
  Interventions: Behavioral: Moderate-intensity continuous training (MCT); Behavioral: Resistance training
- Moderate-intensity continuous training + resistance training + weight loss (Experimental): Tailored moderate-intensity exercise training videos with weekly virtual meetings with a coach + tailored resistance training videos + initiation/intensification of pharmacological weight loss
  Interventions: Behavioral: Moderate-intensity continuous training (MCT); Behavioral: Resistance training; Drug: Weight loss

INTERVENTIONS:
Behavioral: Moderate-intensity continuous training (MCT) — Tailored moderate-intensity exercise training video with weekly virtual meetings with a coach
Behavioral: Resistance training — Resistance training videos assigned to patient
  Arms: Moderate-intensity continuous training + resistance training; Moderate-intensity continuous training + resistance training + weight loss
Drug: Weight loss — Initiation/intensification of weight loss medications, such as semaglutide or tirzepatide
  Arms: Moderate-intensity continuous training + resistance training + weight loss; Moderate-intensity continuous training + weight loss

SUMMARY:
Heart failure with preserved ejection fraction (HFpEF) is associated with a high morbidity and mortality burden. There are limited pharmacological options available for the treatment of HFpEF. Exercise intolerance (EI) is the cardinal symptom of HFpEF, which manifests as dyspnea and fatigue. EI leads to functional deconditioning and reduced quality of life (QOL), both of which elevate risk of death and hospitalization in patients with HFpEF. Supervised exercised training is associated with improvements in exercise capacity and QOL in adults with HFpEF. However, supervised exercise has not been widely utilized for the treatment of HFpEF due to logistical and fiscal barriers.

This study will investigate the effects of a remote exercise training intervention on exercise capacity and skeletal muscle composition in patients with HFpEF, or those at risk for it. In addition, it will compare four different lifestyle interventions for their effects on exercise capacity.

DETAILED DESCRIPTION:
Heart failure (HF) portends substantial morbidity, mortality, and health care costs in the United States and the prevalence of heart failure with preserved ejection fraction (HFpEF) relative to HF with reduced ejection fraction (HFrEF) has been increasing. HFpEF is associated with a high morbidity and mortality burden. There are limited pharmacological options available for the treatment of HFpEF. It is now recognized as a systemic, multi-organ, geriatric syndrome, with exercise intolerance (EI) and functional impairment as the key clinical manifestations. EI leads to functional deconditioning and reduced quality of life (QOL), both of which elevate risk of death and hospitalization in patients with HFpEF. Supervised exercised training is associated with improvements in exercise capacity and QOL in adults with HFpEF. However, supervised exercise has not been widely utilized for the treatment of HFpEF due to logistical and fiscal barriers.

This study will investigate the effects of a remote exercise training intervention on exercise capacity and skeletal muscle composition in patients with HFpEF, or those at risk for it. In addition, it will compare the effects of four different lifestyle interventions on exercise capacity.

The study will be carried out in two phases. In Phase I, 120 participants will undergo three months of home-based moderate-intensity continuous training (MCT), using tailored exercise videos on a mobile or tablet. Participants will also have weekly virtual meetings with a coach to discuss their progress. This will be followed by 3 months of no intervention, to assess the effects of detraining.

In Phase II (at the 6-month mark), 100 participants will be randomized to one of four extended training strategies for 3 months -(i) MCT alone; (ii) MCT plus resistance training; (iii) MCT plus weight loss, or (iv) MCT plus resistance training and weight loss.

The co-primary outcomes are (1) peak VO2, and (2) short physical performance battery score. In addition, participants will undergo CT chest/abdomen/pelvis at 3 months and 6 months to assess change in skeletal muscle composition with MCT

ELIGIBILITY:
Inclusion Criteria:

1. Age>= 18 yrs
2. LVEF (Left Ventricular Ejection Fraction) >= 50%
3. History of HFpEF or at risk of HFpEF

   1. HFpEF diagnosis based on:- -HF hospitalization within 12 months-

      * NT-proBNP >360 pg/mL
   2. Risk of HFpEF based on:-

      * >2 risk factors (h/o diabetes, hypertension, obesity, physical inactivity by self-report)
4. SPPB < 10 or VO2<60th percentile
5. BMI >=28 (for randomization in phase II)
6. Able to use cell phone and mobile application

Exclusion Criteria:

1. Hospitalization 1 month prior to baseline visit
2. History of recurrent falls
3. eGFR (Estimated Glomerular Filtration Rate) <20ml/min/1.73m
4. Active changes in HF therapies over 2 weeks prior to baseline visit
5. Inability participate in exercise training therapy
6. Inability to perform CPET (Cardiopulmonary Exercise Testing) testing
7. Severe left side valvular heart disease
8. End stage pulmonary disease, requiring continuous supplemental oxygen
9. Major surgery within 3 months of screening or major elective surgery during the duration of the study.
10. Unstable weight defined by >5% change in body weight in last 30 days before first study visit.
11. Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-02-18 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Peak Exercise Oxygen Uptake (VO2peak) | Baseline, 3months, 6months, and 9months
  VO2peak indexed to body weight (mL/kg/min) will be the co-primary outcome for the trial. VO2peak is a gold-standard measure of aerobic exercise capacity and will be measured by maximal exercise test using a previously established ergometer protocol
Short Physical Performance Battery (SPPB) | Baseline, 3months, 6months, and 9months
  SPPB will be a co-primary outcome for the trial. Score ranges from 0 to 12, with 0 indicating the worst performance and 12 indicating the best.

SECONDARY OUTCOMES:
Kansas City Cardiomyopathy Questionnaire 12 (KCCQ-12) | Baseline, 3months, 6months, and 9months
  Health-related quality of life will be assessed using the KCCQ-12 questionnaire. This is a self-administered questionnaire that assesses a patient's perception of their heart failure with regard to the psychological, physical, and socioeconomic aspects of life. Scores range from 0 to 100, where 0 indicates the worst possible health status and 100 indicates the best.
6 Minute Walk Distance (6MWD) | Baseline, 3months, 6months, and 9months
  6MWD is a simple and well-validated measure of submaximal exercise capacity and does not require any exercise equipment or advanced training for technicians
General Quality of Life - EQ-5D-5L | Baseline, 3months, 6months, and 9months
  Change in general health-related quality of life assessed using the EuroQol 5 Dimension 5 Level (EQ-5D-5L) instrument. The EQ-5D-5L uses a descriptive system to measure health-related quality of life across five key dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension is rated on five levels of severity-ranging from no problems (Level 1) to extreme problems or inability to function (Level 5). A respondent's answers generate a five-digit health state profile that reflects their unique combination of responses (e.g., 12345), representing one of 3,125 possible health states. This descriptive system enables consistent and standardized assessment of an individual's health status.
Thirty Second Chair Test | Baseline, 3months, 6months, and 9months
  The 30-second chair stand test measures lower-body strength and endurance by counting how many times a person can stand up from a chair and sit down within 30 seconds.
Fried Frailty Phenotype | Baseline, 3months, 6months, and 9months
  The Fried frailty phenotype defines frailty based on five criteria-unintentional weight loss, exhaustion, weakness, slow walking speed, and low physical activity. Each criterion met adds one point to the total score. The Fried Frailty scale has a score range of 0 to 5. A score of 0 means the person is robust or not frail, a score of 1 or 2 indicates pre-frailty (intermediate risk), and a score of 3 or more means the person is considered frail.
Resting cardiac output | Baseline, 3months, 6months, and 9months
  Assess with echocardiography to measure stroke volume and heart rate during rest
Exercise cardiac output | Baseline, 3months, 6months, and 9months
  Assess with echocardiography to measure stroke volume and heart rate responses with graded physical stress.
Intramyocellular fat | Baseline, 3months, 6months, and 9months
  Assessed with non-contrast CT scans of the chest, abdomen, and pelvis. These scans will be used to measure the radiodensity of muscle tissue, quantified in Hounsfield Units (HU). Skeletal muscle tissue is assigned a range of HU values (-29 to +150). Higher fat content lowers the overall muscle density, resulting in lower HU values
Intermuscular Adipose Tissue (IMAT) | Baseline, 3months, 6months, and 9months
  Assessed with non-contrast CT scans of the chest, abdomen, and pelvis. These scans quantify intermuscular adipose tissue (IMAT) using the Hounsfield unit (HU) scale, where IMAT is classified as fat density within a range of -250 to -30 HU. The area of fat deposits is then quantified in square centimeters (cm^2)
Subcutaneous adiposity deposits | Baseline, 3months, 6months, and 9months
  Assessed with non-contrast CT scans of the chest, abdomen, and pelvis. These scans quantify fat deposits using the Hounsfield unit (HU) scale, where fat is defined as a density within a range of -250 to -30 HU. The area of fat deposits is then quantified in square centimeters (cm^2)
Visceral Adiposity Deposits | Baseline, 3months, 6months, and 9months
  Assessed with non-contrast CT scans of the chest, abdomen, and pelvis. These scans quantify fat deposits using the Hounsfield unit (HU) scale, where fat is defined as a density within a range of -250 to -30 HU. The area of fat deposits is then quantified in square centimeters (cm^2)
Pericardial Adiposity Deposits | Baseline, 3months, 6months, and 9months
  Assessed with non-contrast CT scans of the chest, abdomen, and pelvis. These scans quantify fat deposits using the Hounsfield unit (HU) scale, where fat is defined as a density within a range of -250 to -30 HU. The area of fat deposits is then quantified in square centimeters (cm^2)
Lower Body Adiposity Deposits | Baseline, 3months, 6months, and 9months
  Assessed with non-contrast CT scans of the chest, abdomen, and pelvis. These scans quantify fat deposits using the Hounsfield unit (HU) scale, where fat is defined as a density within a range of -250 to -30 HU. The area of fat deposits is then quantified in square centimeters (cm^2)
E/e': Ratio of early mitral inflow velocity (E) to early diastolic mitral annular velocity (e') | Baseline, 3months, 6months, and 9months
  Exercise echocardiography to measure E/e' ratio to assess left ventricular filling pressures at rest and during graded physical stress
Left atrial reservoir strain | Baseline, 3months, 6months, and 9months
  Assessed using echocardiography at rest and during graded physical stress
Left ventricular global longitudinal strain (LV GLS) | Baseline, 3months, 6months, and 9months
  Assessed using echocardiography at rest and during graded physical stress
GAD 7 score | Baseline, 3months, 6months, and 9months
  Change in anxiety symptoms assessed using the Generalized Anxiety Disorder-7 (GAD-7) scale. Total scores range from 0 to 21, with higher scores indicating more severe anxiety symptoms.
PHQ 9 score | Baseline, 3months, 6months, and 9months
  This is a self-administered questionnaire that assesses the severity of depressive symptoms. The PHQ-9 (Patient Health Questionnaire-9) ranges from 0 to 27, with higher scores indicating more severe depressive symptoms.
NT-proBNP | Baseline, 3months, 6months, and 9months
  Serum level of NT-proBNP (N-terminal pro-brain natriuretic peptide), a biomarker that reflects cardiac stress.
High-sensitivity troponin I | Baseline, 3months, 6months, and 9months
  Serum high-sensitivity troponin I reflects ongoing low-grade myocardial injury and is a marker of disease severity and prognosis in chronic heart failure.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States